CLINICAL TRIAL: NCT07274449
Title: Exploratory Clinical Study on Memory NK Cell Therapy for Advanced Metastatic Solid Tumors
Acronym: NK
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC2025-0001-02
Record Dates: First submitted 2025-11-17; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Memory NK Cell Therapy
  Interventions: Biological: Memory-Like NK Cells

INTERVENTIONS:
Biological: Memory-Like NK Cells — The study employs iRGD-modified cytokine-induced memory-like NK cells. These memory NK cells-primed with IL-12, IL-15, and IL-18-exhibit enhanced antitumor functionality, characterized by ↓KIR expression, ↑NKP30 expression, increased IFN-γ/TNF-α secretion, and significantly improved in vitro cytotoxicity. The iRGD modification, applied to cell membranes using our proprietary tumor-penetrating peptide technology, confers active tumor-targeting and tissue-penetrating capabilities to the NK cells.

SUMMARY:
This study is a single-center, prospective, Phase Ib/II clinical trial designed to evaluate the safety and efficacy of cell membrane-modified memory NK cells in treating patients with advanced metastatic solid tumors.

The primary objective of this study is to evaluate the safety and tolerability profile of memory NK cells administered in combination with standard therapy in the Intent-to-Treat (ITT) population. The assessment will be based on the following endpoints: 1）Incidence of dose-limiting toxicities (DLTs)； 2) Frequency and severity of adverse events; 3) Occurrence of clinically significant abnormalities in laboratory parameters, physical examinations, and vital signs.

The secondary Study Objectives: 1) To evaluate the preliminary efficacy of the combination regimen by assessing the objective response rate (ORR), duration of response (DOR), progression-free survival (PFS), overall survival (OS), and serial changes in tumor markers; 2) To characterize the pharmacokinetic profile of memory NK cells when used in combination with standard therapy within the ITT population.

A pilot cohort of 6 patients will first be enrolled to assess the safety of NK cell therapy, with dose-limiting toxicities (DLT) evaluated over a 21-day observation period following the last NK cell infusion. If safety is confirmed, a protocol amendment for cohort expansion will be submitted to the Ethics Committee.

DETAILED DESCRIPTION:
After passing screening, eligible subjects will have haploidentical mononuclear cells collected for memory NK cell culture. When the cell count reaches the specified 5×10^9/L after approximately 2-3 weeks of culture, cell reinfusion will be initiated. Each cycle consists of three reinfusions (on Days 1, 8, and 15). Standard guideline-recommended therapy will be administered 3-5 days before the first reinfusion of each cycle. One day prior to each reinfusion, a 2Gy low-dose immunotherapeutic radiation may be administered to tumor-involved lesions based on the patient's performance status. Efficacy will be evaluated after two cycles of reinfusion. For patients with rapid tumor progression or high tumor burden, investigators may administer standard chemotherapy during the cell culture phase based on the patient's condition. Subsequently, subjects will continue maintenance therapy according to the original standard treatment until any of the following occurs: disease progression, intolerable toxicity, initiation of new antitumor therapy, withdrawal of informed consent, loss to follow-up, death, or other protocol-specified conditions for treatment discontinuation, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* The study participants are able to understand the informed consent form, voluntarily participate and sign the informed consent form.
* The study participant is 18 ~ 75 years old on the day of signing the informed consent.
* The Eastern Cooperative Oncology Group (ECOG) performance status score (ECOG) is 0-3, which allows bed rest most of the time, but can still maintain the minimum daily self-care ability.
* Estimated survival time>=8 weeks.
* Patients with solid tumors such as colorectal cancer, gastric cancer, lung cancer, ovarian cancer, and neuroendocrine tumors who have failed first-line standard therapy recommended by the guidelines (disease progression after treatment or intolerable toxic side effects of treatment) should have at least one measurable lesion for efficacy evaluation.
* All research participants should provide archived or freshly obtained tumor tissue samples or 5 unstained tumor tissue section samples within 2 years before signing the informed information as much as possible, and newly obtained tumor tissue samples are preferred. The patient's tumor tissue was stained by immunohistochemistry, and 40% of the tumor cell membrane was stained with (2/3) at least one of the targets of integrin aVβ3, CLDN6, KKLC-1, DLL3, and mesothelin.
* The patient has adequate organ and bone marrow function, defined as follows: Complete blood count: white blood cell count >=2.0×10^9/L, neutrophil count >=1.0×10^9/L, hemoglobin >=7.0g/dL, platelet count >=75×10^9/L; Liver function: total bilirubin <=1.5× upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) in study participants without liver metastases<=2.5×ULN. There are liver metastases study participants requested: ALT and AST <=5×ULN. Renal function: serum creatinine (Scr) <=1.5×ULN. Adequate coagulation: defined as international normalized ratio (INR) <=1.5 or prothrombin time (PT) <=1.5 times ULN; If the study participant is receiving anticoagulant therapy, as long as the PT is within the intended range of the anticoagulant medication.
* Patients of childbearing age need to take appropriate protective measures (contraceptive measures or) before enrollment and during the test other methods of birth control).
* Have signed the informed consent form and be able to comply with the visit and related procedures specified in the program.

Exclusion Criteria:

* Palliative local therapy targeting lesions within 2 weeks prior to the first dose; systemic non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin) within 2 weeks prior to the first dose; use of herbal or traditional Chinese medicines with anti-tumor indications within 2 weeks prior to the first dose.
* History of other malignancies, except for carcinoma in situ of the cervix, treated squamous cell carcinoma or urothelial bladder tumors (Ta and TIS), or other malignancies that have undergone curative therapy (at least 5 years prior to enrollment).
* Uncontrolled comorbid conditions, including but not limited to active bacterial/fungal infections, symptomatic congestive heart failure, unstable angina, or arrhythmias.
* Concurrent HIV infection, active hepatitis B (HBV DNA >=500 IU/mL), or hepatitis C.
* Uncontrolled coronary artery disease, asthma, cerebrovascular disease, or other conditions deemed ineligible by the investigator.
* Poorly controlled comorbidities, including active infections, congestive heart failure, unstable angina, arrhythmias, or congenital long QT syndrome; corrected QTc interval >500 ms (Fridericia's formula) at screening.
* Subjects with autoimmune diseases or immunodeficiency disorders.
* Use of immunosuppressive drugs within 4 weeks prior to the first dose, excluding: a) Intranasal inhaled corticosteroids or local steroid injections (e.g., intra-articular); b) Systemic corticosteroids ≤10 mg/day prednisone equivalents; c) Corticosteroids as premedication for hypersensitivity (e.g., pre-CT contrast).
* Subjects requiring chronic systemic corticosteroids or other immunosuppressive agents (excluding inhaled corticosteroids).
* Administration of live attenuated vaccines within 4 weeks prior to the first dose or planned during the study.
* Major surgery (e.g., craniotomy, thoracotomy, laparotomy) within 4 weeks prior to the first dose or anticipated need for major surgery during the study.
* History of gastrointestinal perforation/fistula, bowel obstruction (including incomplete obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within 6 months prior to enrollment.
* Gastrointestinal bleeding or high bleeding risk within 2 weeks prior to enrollment.
* Symptomatic central nervous system metastases requiring clinical intervention.
* Pregnancy or lactation.
* Known hypersensitivity to the investigational drug or its excipients.
* Subjects unable to undergo immunotherapy due to social or geographical factors.
* Any unresolved condition that may compromise safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to one year.

SECONDARY OUTCOMES:
Overall Survival | From clinical trial enrollment until the date of death from any cause, assessed up to one year.
Disease control rate | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to one year.
Duration of control | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to one year.
Objective response rate | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to one year.
Progression free survival | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No